CLINICAL TRIAL: NCT02835469
Title: Non-Interventional Clinical Study on Efficacy and Safety of Highly Purified Human Menopausal Gonadotrophin (HP-hMG) Menopur® Multidose in Korean Female Patients With Infertility
Brief Title: A Study on Efficacy and Safety of Menopur® Multidose in Korean Female Patients With Infertility
Status: Completed | Type: Observational
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 000258
Record Dates: First submitted 2016-06-28; First posted 2016-07-18 (Estimated); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Menotropins

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Menopur® Multidose: Treatment according to routine clinical practice.
  Interventions: Drug: Menotrophin

INTERVENTIONS:
Drug: Menotrophin
  Other Names: Menopur® Multidose

SUMMARY:
The purpose of this study is to investigate the ongoing pregnancy rates at 10-11 weeks after embryo transfer in patients treated with Menopur® Multidose

ELIGIBILITY:
Inclusion Criteria:

* Decision made to prescribe Menopur® multidose according to Summary of product characteristics
* The study cycle will be either

  * 1st controlled ovarian stimulation cycle ever, or
  * 2nd controlled ovarian stimulation cycle ever, or
  * 1st or 2nd controlled ovarian stimulation cycle after having achieved ongoing pregnancy in a previous controlled ovarian stimulation cycle (note: the subject cannot be included if she has had made more than one failed cycle before the cycle resulting in ongoing pregnancy)

Exclusion Criteria:

* Known ovarian disease (e.g. ovarian cysts, polycystic ovarian disease etc.)
* Diagnosed as "poor responder", defined as either

  * >20 days of gonadotrophin stimulation in a previous controlled ovarian stimulation cycle, or
  * any previous cancellation of a controlled ovarian stimulation cycle due to limited follicular response, or
  * development of less than 4 follicles ≥15 mm in a previous controlled ovarian stimulation cycle
* Ovarian hyperstimulation syndrome (OHSS)

Ages: 19 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Fertility clinics
Sampling Method: Non-Probability Sample
Enrollment: 412 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Ongoing pregnancy rate | 10-11 weeks after embryo transfer
  Defined as presence of at least 1 intrauterine pregnancy with a viable fetus

SECONDARY OUTCOMES:
Mean Follicle Stimulating Hormone (FSH) level | At baseline and last stimulation day (max 20 days after start of stimulation)
Mean Luteinizing Hormone (LH) level | At baseline and last stimulation day (max 20 days after start of stimulation)
Mean Estradiol 2 (E2) level | At baseline and last stimulation day (max 20 days after start of stimulation)
Mean endometrial thickness | On last stimulation day (max 20 days after start of stimulation)
  Measured by transvaginal ultrasound
Follicular development | On last stimulation day (max 20 days after start of stimulation)
  Number and size of follicles measured by transvaginal ultrasound
Number of oocytes retrieved | 36 hours (±2h) after human Chorionic Gonadotrophin (hCG) administration
Fertilization rate | 1 day after oocyte retrieval
  Number of oocytes with 2 pronuclei divided by number of metaphase II oocytes

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (1):
- CL Hospital (there may be other sites in this country), Gwangju, South Korea